CLINICAL TRIAL: NCT06848686
Title: Prevention Ambassadors: an HIV Self-testing Intervention to Promote HIV Service Engagement in the Networks of SSP Clients
Brief Title: Prevention Ambassadors: Intervention to Promote HIV Service Engagement in the Networks of SSP Clients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of California, San Diego (Other); University of California, Riverside (Other); Dap Health (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-2023-0051; R34DA058389 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention Ambassadors (Experimental)
  Interventions: Behavioral: Prevention Ambassadors
- SSP Standard of Care (Other)
  Interventions: Behavioral: SSP Standard of Care

INTERVENTIONS:
Behavioral: Prevention Ambassadors — Delivery of prevention supplies and information on local services plus training to build the capacity of PWUD to distribute HIV self-testing (HIVST) kits with information and referrals to other PWUD in their social networks to promote HIV testing and HIV service engagement among PWUD.
  Arms: Prevention Ambassadors
Behavioral: SSP Standard of Care — Delivery of prevention supplies and information on local services.
  Arms: SSP Standard of Care

SUMMARY:
HIV testing and service uptake are infrequent among people who use drugs (PWUD) in the United States. In partnership with a community-based syringe service program (SSP), this project will develop the SSP-based "Prevention Ambassadors" (PA) intervention to promote HIV testing and service uptake among PWUD via the secondary distribution (i.e., peer delivery) of HIV self-testing (HIVST) kits with local HIV service information and referrals to HIV service navigation in the social networks of SSP clients (i.e., PWUD). The PA intervention will then be piloted to assess its preliminary effects, acceptability, and feasibility among PWUD in the Ending the HIV Epidemic priority jurisdiction of Riverside County, California.

ELIGIBILITY:
Index Participant Inclusion Criteria:

* Being greater than or equal to 18 years old
* Reporting drug use (past month)
* Having other people who use drugs (PWUD) in one's social network
* Being willing to talk about HIV testing and services with at least 2 PWUD in their networks and attempt to refer them to the study
* Speaking English fluently

Peer-Recruit Participant Inclusion Criteria:

* Being greater than or equal to 18 years old
* Reporting drug use (past 3 months)
* Being recruited by an index participant (evidenced by presenting the coupon used to recruit them)
* Speaking English fluently

Exclusion Criteria:

- Persons who participated in formative study activities related to the development of the PA intervention will not be eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
HIV testing (past 3 months) | 3-month follow-up
  Self-reported via survey and abstracted from medical record
Linkage to PrEP/HIV care (past 3 months) | 3-month follow-up
  Self-reported via survey and abstracted from medical record
PrEP/ART uptake (past 3 months) | 3-month follow-up
  Self-reported via survey and abstracted from medical record

SECONDARY OUTCOMES:
PA Acceptability (Peer-Recruit Participants) | Baseline
  Self-reported via survey
PA Acceptability (Index Participants) | 3-month follow-up
  Self-reported via survey
PA Feasibility (Peer-Recruit Participants) | Baseline
  Self-reported via survey
PA Feasibility (Index Participants) | 3-month follow-up
  Self-reported via survey

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Pines, Principal Investigator — San Diego State University; Angela R Bazzi, Principal Investigator — University of California, San Diego
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon review of written requests from researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Approximately 6 months after the publication of the study's primary findings.
Access Criteria: Requests from researchers for de-identified data will be reviewed by the research team (Multiple Principal Investigators and Co-Investigators).